CLINICAL TRIAL: NCT04725877
Title: A Phase 1a, Randomized, Placebo-Controlled Study to Evaluate the Safety and Immunogenicity of a Prototype Human CMV-based Vaccine for Human Immunodeficiency Virus (HIV) in Healthy Volunteers
Brief Title: VIR-1111: A Prototype Human CMV-based Vaccine for Human Immunodeficiency Virus (HIV) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vir Biotechnology, Inc. (Industry)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VIR-1111-2001
Record Dates: First submitted 2021-01-08; First posted 2021-01-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: HIV I Infection
Keywords: HIV; Vaccine; CMV; Cytomegalovirus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VIR-1111 (Experimental)
  Interventions: Biological: VIR-1111
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: VIR-1111 — VIR-1111 is administered as a 1 mL subcutaneous injection in the deltoid area of the upper arm on Day 1 and Day 57.
  Arms: VIR-1111
Drug: Placebo — A placebo (Tris NaCl Sucrose formulation buffer) given by subcutaneous injection.
  Arms: Placebo

SUMMARY:
This is a Phase 1a, first in human study in which healthy adult participants who are considered to be at low-risk for HIV infection and are seropositive for cytomegalovirus (CMV) will receive two doses of VIR-1111 or placebo. These participants will be assessed for safety, reactogenicity, tolerability and immunogenicity. There is an optional long-term follow-up study that would lengthen study participation for up to 3 years post-first dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or healthy females of non-child-bearing potential between the ages of 18 to 50 at the time of screening
* Positive CMV serostatus
* Assessed by clinic staff as being low risk for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last protocol visit
* Willing to use condoms during intercourse through Week 36 or the end of the study
* Willing to undergo HIV testing, risk reduction counseling, and receive HIV test results
* Willing to comply with the protocol requirements regarding donation of blood, sperm or other tissues
* In the opinion of the Investigator, generally in good health as determined from medical history and no clinically significant findings from physical examinations, vital signs, and laboratory values

Exclusion Criteria:

* Live in a home with children under the age of 6
* Routine provision of child care to children under the age of 6
* Have close contact with immunocompromised individuals
* Have close contact with pregnant women or a partner planning to become pregnant during the course of the study
* Health care provider who routinely comes into contact with immunosuppressed patients or pregnant women
* Participant is immunocompromised
* Participant has an autoimmune disorder
* Positive HIV test at the time of study screening
* Receipt of another investigational HIV or CMV vaccine candidate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with any treatment-emergent adverse events (AEs) | Day 1 through 36 weeks
  A treatment-emergent AE is any AE with an onset date on or after the investigational product start date and no later than 36 weeks after permanent discontinuation of the investigational product.
Number of participants with any serious AEs (SAEs) | Day 1 through 36 weeks
  An SAE is any life-threatening event or one that results in hospitalization, significant disability/incapacity, death or congenital anomaly/birth defect.
Number of participants with any local site reactogenicity event after first dose | Day 1 through 14 days after first dose
  Signs and symptoms will be captured at the injection site (e.g., pain/tenderness, swelling, redness and induration) through self-assessment via participant diaries and in-person clinical assessments.
Number of participants with any local site reactogenicity event after second dose | Day 1 through 14 days after second dose
  Signs and symptoms will be captured at the injection site (e.g., pain/tenderness, swelling, redness and induration) through self-assessment via participant diaries and in-person clinical assessments.
Number of participants with any systemic reactogenicity event after first dose | Day 1 through 14 days after first dose
  Systemic signs and symptoms (fever, headache, fatigue, arthralgia, myalgia, malaise, nausea, vomiting or chills) through self-assessment via participant diaries and in-person clinical assessments.
Number of participants with any systemic reactogenicity event after second dose | Day 1 through 14 days after second dose
  Systemic signs and symptoms (fever, headache, fatigue, arthralgia, myalgia, malaise, nausea, vomiting or chills) through self-assessment via participant diaries and in-person clinical assessments.
Number of participants with any treatment-emergent clinical laboratory abnormalities (chemistry, hematology and liver function tests) | Day 1 through 36 weeks
  A treatment-emergent clinical laboratory abnormality is a clinical laboratory value that increases at least 1 toxicity grade from baseline at any postbaseline timepoint up to 30 days after permanent discontinuation of study drug. Clinical laboratory abnormalities are graded using DAIDS Table for Grading and Severity of Adult and Pediatric Events, Corrected Version 2.1, July 2017.
Number of participants with CMV vector viremia (blood) | Day 1 through 36 weeks
  Quantitative polymerase chain reaction (qPCR) for CMV will be performed on participant blood samples collected throughout the study. Positive samples will undergo follow-up confirmatory PCR testing to differentiate wild-type CMV from CMV vaccine vector sequences.
Number of participants with CMV vector shedding (urine and saliva) | Day 1 through 36 weeks
  Quantitative polymerase chain reaction (qPCR) for CMV will be performed on both saliva and urine samples collected from participants throughout the study to monitor for viral shedding. Positive samples will undergo follow-up confirmatory PCR testing to differentiate wild-type CMV from CMV vaccine vector sequences.

SECONDARY OUTCOMES:
Frequency of CMV-specific CD8 T cells via peptide stimulation, intracellular cytokine staining and flow cytometry to detect IL-2 AND/OR IFNg AND/OR TNFa | 0-36 weeks
Frequency of CMV-specific CD4 T cells via peptide stimulation, intracellular cytokine staining and flow cytometry to detect IL-2 AND/OR IFNg AND/OR CD154 | 0-36 weeks
Frequency of HIV-1 Clade A Gag-specific CD4 T cells via peptide stimulation, intracellular cytokine staining and flow cytometry to detect IL-2 AND/OR IFNg AND/OR TNFa AND/OR CD154 | 0-36 weeks
Frequency of HIV-1 Clade A Gag-specific CD8 T cells T cells via peptide stimulation, intracellular cytokine staining and flow cytometry to detect IL-2 AND/OR IFNg AND/OR TNFa | 0-36 weeks
Memory phenotype of CMV-specific CD4 T cells via flow cytometry analysis of CD45RA, CCR7, CD27, CD28 AND/OR CD95. | 0-36 weeks
Memory phenotype of CMV-specific CD8 T cells via flow cytometry analysis of CD45RA, CCR7, CD27, CD28 AND/OR CD95 | 0-36 weeks
Memory phenotype of HIV-1 Clade A Gag-specific CD4 T cells via flow cytometry analysis of CD45RA, CCR7, CD27, CD28 AND/OR CD95 | 0-36 weeks
Memory phenotype of HIV-1 Clade A Gag-specific CD8 T cells via flow cytometry analysis of CD45RA, CCR7, CD27, CD28 AND/OR CD95 | 0-36 weeks
Binding titers of CMV-specific IgG antibodies | 0-36 weeks
Binding titers of HIV Clade A Gag-specific IgG antibodies | 0-36 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Investigative Site, Miami, Florida
  - Investigative Site, Seattle, Washington
  - Investigative Site, Madison, Wisconsin